CLINICAL TRIAL: NCT07055412
Title: To Evaluate the Pharmacokinetics and Safety of Y-3 for Injection in Patients With Hepatic Insufficiency and Healthy Subjects
Brief Title: Y-3 for Injection in Patients With Hepatic Insufficiency and Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Y-3-LC-07
Record Dates: First submitted 2025-06-20; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pharmacokinetic Differences; Y-3; Saftey; Mild Hepatic Insufficiency; Moderate Hepatic Insufficiency; Normal Hepatic Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Y-3（40mg） (Experimental)
  Interventions: Drug: Y-3 for injection（40mg）

INTERVENTIONS:
Drug: Y-3 for injection（40mg） — The investigational drug (Y-3) consists of two parts: Y-3 for injection (lyophilized powder) and Solvent for Y-3 for injection (concentrated solution).
  Name: Y-3 for injection Strength: 20 mg Dosage Form: Lyophilized powder for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd. Name: Reconstitution diluent for Y-3 for injection Strength: 3ml (containing 0.6 g propylene glycol) Dosage Form: Concentrated solution for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd.

SUMMARY:
The goal of this clinical trial is to assess the pharmacokinetic profiles and safety of Y-3 in subjects with mild hepatic insufficiency (Child-Pugh: grade A), moderate hepatic insufficiency (Child-Pugh: grade B) and gender, age, and weight matching normal hepatic function, so as to provide a scientific basis for rational clinical medication in patients with hepatic insufficiency.

The main questions it aims to answer are:

What the pharmacokinetic profiles of Y-3 (40 mg ) in subjects with mild hepatic insufficiency (Child-Pugh: grade A), moderate hepatic insufficiency (Child-Pugh: grade B) and gender, age, and weight matching normal hepatic function？ If drug Y-3 (40mg ) is safe and tolerate in subjects with mild hepatic insufficiency (Child-Pugh: grade A), moderate hepatic insufficiency (Child-Pugh: grade B) and gender, age, and weight matching normal hepatic function.

Investigators will compare pharmacokinetic safety profiles of Y-3 (40 mg ) in subjects with different hepatic functions( mild hepatic insufficiency, moderate hepatic insufficiency, normal.

Participants will:

Take drug Y-3 (40 mg) only once. Answer questions regarding your medical history. Comply with the study procedures and requests. Complete all tests and collections of PK Sampling. Fasting for more than 10 hours before administration, water abstinence for 1 h before and after administration, and eating standard lunch and dinner 4 hours and 10 hours after starting administration.

Must not use of nicotine-containing products (including nicotine patches). Must not do strenuous exercise for 1 hour before each clinical laboratory test blood draw. Subjects may engage in light recreational activities for the duration of the study.

Follow your doctor's instructions, answer the investigator's questions about your health status truthfully, and cooperate with the test-related tests.

During the experiment, the test should be completed in strict accordance with the requirements of the investigator, and the test-related work such as drug administration and sample collection should be conscientiously cooperated, and the research center should not leave the research center without authorization, and the rules and regulations of the research center and the investigator 's propaganda and education should be observed. Any medication taken should be reported truthfully.

Must come to the hospital at the agreed follow-up time with the investigator and you.

Inform the investigator or relevant person about any changes in your health status, including any favorable or unfavorable changes.

Must not participate in any other drug clinical trials during this trial. Must tell your investigator about all medical treatments you plan to receive during the study, such as elective surgery or radiation therapy.

In addition to yourself, at least one member of your family is expected to be aware of the clinical research you will be involved in and care about your health, and will be able to provide feedback to your doctor about your health during follow-up visits. Your family should promptly notify your study physician if you become seriously unwell, including hospitalization for treatment.

Notify your investigator if your address, phone number, or other contact information changes.

Must not use medications that may interfere with PK or safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria for inclusion:

  1. The subject fully understands the purpose and requirements of this trial, voluntarily participates in the clinical trial and signs a written ICF, strictly abide by the clinical study protocols and requirements to complete the whole study process;
  2. Be 18~70 years old (including the boundary value) on the day of signing the ICF, both male and female;
  3. At screening, the weight of male subjects ≥ 50kg, the weight of female subjects ≥ 45kg, and the body mass index [BMI=Weight (kg)/height 2 (m2)] within the range of 18.0~30.0kg/m2 (including boundary value);
  4. Subjects (including their spouses or partners) have no sperm or egg donation programs, no fertility plans, and voluntary strict contraceptive use during the trial and within 3 months after the completion of the trial, see Appendix 1: Contraceptive measures administration and contraceptive requirements;
  5. The estimated glomerular filtration rate (eGFR) calculated using the modification of diet in renal disease (MDRD) formula ≥ 80 ml/min/1.73 m2. (See Appendix 2: Glomerular Filtration Rate Calculation Formula);

     Subjects with hepatic insufficiency must also meet all of the following criteria:
  6. Chronic liver injury caused by primary liver disease (such as hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, non-alcoholic liver disease, fatty liver, etc.) or clinical diagnosis of liver cirrhosis (see Appendix 3: Diagnostic Criteria for Liver Cirrhosis) caused by primary liver disease, Child-Pugh grade A or B patients with hepatic insufficiency (see Appendix 4: Liver Function Assessment for Child-Pugh classification), and have not used albumin within 14 days before screening, and the investigator judged that patients with mild hepatic insufficiency need to be clinically stable ≥for 28 days before taking the investigational products, and patients with moderate hepatic insufficiency need to be clinically ≥stable for 14 days before taking the investigational products, and the investigator judges that the subject's liver function status is stable from 2 weeks before screening to the end of the study, and no obvious deterioration will occur;
  7. Have not taken any medication within 1 week before screening; or those who require long-term treatment for liver damage, complications and/or other concomitant diseases should have stable medication for at least 4 weeks (stable medication is judged by the investigator, except for drugs prohibited by the protocol).

     Subjects with normal liver function also need to meet all of the following criteria:
  8. The demographic mean of subjects in the normal hepatic function group (Group C) at screening must meet the following matching standard:

     1. Sex matching with liver insufficiency group (group A and group B), with a mean value of ±1 case;
     2. Age matching with hepatic insufficiency group (Group A and Group B) with a mean ± 10 years;
     3. Body weight matching with hepatic insufficiency group (group A and group B) with a mean of ±10%.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible for inclusion in this study:

  1. Irritable the physique, such as those with a known history of allergy to two or more substances, or those with allergic diseases, or those with a history of allergy to investigational products or excipients (15-hydroxystearate polyethylene glycol, propylene glycol, potassium dibasic phosphate, potassium dibasic phosphate trihydrate, mannitol);
  2. Those who have special dietary requirements and cannot comply with the uniform diet;
  3. Patients with clinically significant ECG abnormalities (tachycardia/bradycardia, II-III degree atrioventricular block or QTcF interval prolongation (QTcF>450ms for males and >470ms for females) (corrected according to Fridericia's formula: QTcF=QT/(RR^0.33), RR=60/heart rate) or other clinically significant abnormalities judged by the investigator to be unsuitable for participating in this study);
  4. Those who have serious infection, trauma, gastrointestinal surgery or other surgical procedures within 4 weeks before screening, or those who plan to undergo surgical treatment during the trial or have a tendency to be hospitalized;
  5. Those who have lost blood or donated ≥ 400 mL of blood within 3 months before dosing, or who have received blood transfusion or used blood products within 1 month, or who plan to donate blood within 1 month after the end of this trial;
  6. Those who have used medium or strong inhibitors or inducers of CYP450 enzyme within 1 month before dosing (such as phenytoin, rifampicin, carbamazepine, fluvoxamine, enoxacin, ticlopidine, gemfibrozil, clopidogrel, clarithromycin, itraconazole, ketoconazole, ritonavir, etc., see Appendix 5: List of Common Drugs for CYP Enzyme Inhibitors or Inducers) or UGT enzyme inhibitors or inducers (such as atazanavir, probenecid, valpendict, mefenamic acid, carbamazepine, rifampicin) within 1 month before dosing , phenytoin, efaviren, phenobarbital, ritonavir, etc., see Appendix 6: List of common drugs for UGT enzyme inhibitors or inducers);
  7. Those who have consumed excessive amounts of tea, coffee and/or caffeinated beverages per day (an average of more than 8 cups per day, 1 cup = 250mL) within 3 months before screening, and those who cannot withdraw during the trial; or those who have consumed a special diet (including dragon fruit, mango, grapefruit, xanthine-rich food, chocolate, etc.) within 2 weeks before screening;
  8. Those who have participated in other clinical trials and received investigational products within 3 months before screening, or those who plan to participate in other clinical trials during this study;
  9. Those who are current or previous alcoholics or regular drinkers within 6 months prior to screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360mL of beer or 45mL of spirits with 40% alcohol or 150mL of wine), or those who have a positive alcohol breath test at baseline (alcohol breath test result >0 mg/100 mL) or those who cannot withdraw during the trial;
  10. Those with a history of drug abuse or drug use or a positive urine drug screen;
  11. Those who are cigarette-addict or smoking more than 5 cigarettes per day within 3 months prior to screening or habitual use of nicotine-containing system and are unable to withdraw during the test;
  12. Those who have received vaccination within 30 days before screening, or plan to be vaccinated during the study;
  13. Pregnant or lactating women, or women of childbearing age who have a positive blood pregnancy test;
  14. Patients who have difficulty in venous blood collection and cannot tolerate venipuncture or fainting needles and blood;
  15. Subjects with poor compliance in the opinion of the investigators, or with other factors that are not suitable for participating in this trial.

      Subjects with hepatic insufficiency who meet any of the following exclusion criteria are excluded:
  16. Subject has any of the following conditions: drug-induced liver injury, history of liver transplantation, acute liver impairment due to various causes, liver failure complicated by infection and/or hepatic encephalopathy, hepatocellular carcinoma;
  17. Patients with liver cirrhosis who are considered inappropriate by the investigator, such as hepatorenal syndrome, active bleeding caused by esophageal and gastric variceal rupture, severe/advanced ascites or pleural effusion requiring puncture and drainage and albumin supplementation;
  18. Patients with primary biliary cirrhosis, biliary obstruction, cholestatic liver disease and other diseases that affect bile excretion;
  19. Laboratory test results consistent with any of the following at screening: (a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5×ULN; (b) Absolute neutrophil value (NE#) < 0.75×109/L; (c) Hemoglobin (HGB) < 80 g/L;(d) Abnormal alpha-fetoprotein (AFP) value (>100ng/mL) requiring liver ultrasonography or other imaging examinations (CT, MRI, etc.), excluding subjects with suspected hepatocellular carcinoma; (e) Platelet < 50×109/L;
  20. Those who are screened positive for HIV antibody and Treponema pallidum specific antibody;
  21. In addition to the primary liver disease itself, those who have suffered from other serious organ system diseases in the past or at present, including but not limited to gastrointestinal, respiratory, renal, neurological, hematologic, endocrine, tumor, immune, psychiatric or cardiovascular and cerebrovascular diseases, which are judged by the research doctor to be unsuitable for participating in this trial;
  22. Those who have used any prescription medicines, over-the-counter medicines, any vitamin products or Chinese herbal medicines other thanmedicines for the treatment of liver insufficiency or their comorbid chronic diseases within 14 days before administration;
  23. Systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg; Pulse < 50 bpm or > 100 bpm;

      Subjects with normal hepatic function who meet any of the following exclusion criteria are excluded:
  24. Those who have a history of liver impairment in the past, or those who have and may have liver impairment as indicated by physical examination and laboratory examination at screening;
  25. Those who have suffered or are currently suffering from any clinical serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, cardiovascular and cerebrovascular, psychiatric and metabolic abnormalities or any other diseases that can interfere with the test results;
  26. Those with abnormal physical examination, vital signs, laboratory tests (Hematology, urine routine, blood biochemistry, coagulation function), 12-lead electrocardiogram, chest X-ray (anterior position), abdominal B-ultrasound (liver, spleen, gallbladder, pancreas, and both kidneys) and other examination abnormalities judged by the investigator to be clinically significant;
  27. Those who test positive for hepatitis B virus surface antigen, hepatitis C virus antibody, HIV antibody, and Treponema pallidum specific antibody;
  28. Have taken any medication (including prescription medicine, over-the-counter medicine, Chinese herbal medicines, vitamins, health products) within 14 days prior to dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Cmax of Y-3 (40 mg ) in subjects with mild hepatic insufficiency , moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin | single-dose administration period (Day1-Day6)
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the AUC 0-t of of Y-3 (40 mg ) in subjects with mild hepatic insufficiency , moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1).
Evaluate the AUC 0-∞ of Y-3 (40 mg) in subjects with mild hepatic insufficiency , moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).

SECONDARY OUTCOMES:
Evaluate the Tmax of Y-3 (40 mg ) in subjects with mild hepatic insufficiency , moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the t1/2 of Y-3 (40 mg ) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Terminal elimination half-life. t1/2 = ln2/λ
Evaluate the λz of Y-3 (40 mg ) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the AUC_%Extrap of Y-3 (40 mg ) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the Vz of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Volume of distribution. Vz = Div/AUC0-∞/λz
Evaluate the CL of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Total body clearance. CLz = Div /AUC0-∞
Evaluate the MRT 0-t of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Mean residence time within the time from time zero to the lowest testing plasma concentration. MRT0-t = AUMC0-t/AUC0-t.
Evaluate the MRT 0-∞ of Y-3 (40 mg ) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by venous blood and Phoenix WinNonlin. | single-dose administration period (Day1-Day6)
  Mean residence time extrapolated from zero to infinity. MRT 0-∞ = AUMC 0-∞/AUC 0-∞.
Evaluate the safety of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic by Incidence of subject getting abnormal results of physical examinations after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Evaluate the safety of Y-3 in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic functionby Incidence of subject getting abnormal results of blood pressure after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. blood pressure will be assessed by electronic sphygmomanometer.
Evaluate the safety of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic functionby Incidence of subject getting abnormal results of respiration after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. respiration will be assessed by nurses.
Evaluate the safety of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic functionby Incidence of subject getting abnormal results of pulse after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. pulse will be assessed by nurses.
Evaluate the safety of Y-3 in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by Incidence of subject getting abnormal results of body temperature after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. body temperature will be assessed by thermometer.
Evaluate the safety of Y-3 (40 mg ) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by Incidence of subject getting abnormal results of 12-lead ECG after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by Incidence of abnormal results of laboratory tests after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of Y-3 (40 mg) in subjects with mild hepatic insufficiency, moderate hepatic insufficiency and gender, age, and weight matching normal hepatic function by the rates of adverse events after treatment. | This study comprises a screening period (Day -28 to Day -1), a baseline period (Day -1), a treatment period (Day1 - Day6), and a safety follow-up period (Day10±1).
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe".
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.

IPD SHARING:
Plan to Share IPD: No